CLINICAL TRIAL: NCT02642328
Title: Effects of Eight Sessions of High Intensity Interval Training (HIIT) With Strength/Power Exercises on VO2Max Gains and Aerobic Performance
Brief Title: High Intensity Interval Training With Strength/Power Exercises on VO2Max
Acronym: Strength
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidade Federal do Rio de Janeiro (Other)
Responsible Party: Principal Investigator, Alberto Souza de Sá Filho, Doctorade in Mental Health, Universidade Federal do Rio de Janeiro
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: UNIG 01
Record Dates: First submitted 2015-12-05; First posted 2015-12-30 (Estimated); Last update posted 2015-12-30 (Estimated); Status verified 2015-12

CONDITIONS: Healthy
Keywords: VO2Max; Aerobic Exercise; Physical Conditioning
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HIIT Training (Experimental): Circuit training with strength and power. The chosen exercises were (random order): Sit-Ups, Mountain Climbers, Plank, Side Skater, Push Ups, Ground Support with Vertical Jump, Overhead Squat, Box Jump.Time total = 4 minutes
  Interventions: Other: Control
- Control (Active Comparator): Running aerobic exercise at 65% of VO2Max
  Interventions: Other: HIIT Training

INTERVENTIONS:
Other: HIIT Training — Circuit of high intensity interval training (HIIT) with Strength and Power Exercises for 4 minutes (20 sec of stimulus / 10 sec rest)
  Other Names: HIIT
  Arms: Control
Other: Control — Continuous aerobic exercise at 65% of VO2Max
  Other Names: Aerobic Exercise
  Arms: HIIT Training

SUMMARY:
Traditionally, strength training and power is the main objective of providing only muscle conditioning, without possible gains on the VO2Max, however, not for aerobic performance.

DETAILED DESCRIPTION:
A total of 10 visits will be performed. The subjects will be divided into two exercise groups: 1) control group (CG) who performed only aerobic activity of running or walking at moderate intensity (65% VO2max); and 2) strength and power exercise group (GFP), which held the protocol circuit. On the first visit the subjects answer an initial questionnaire of risk stratification for coronary artery disease, and performed a maximal aerobic exercise test.

The subjects performed the interval protocol with strength and power exercises at high intensity in circuit. 20 seconds stimuli will be provided with 10 seconds passive recovery, totaling 4 minutes. In the last session the subjects will be performed the same initial procedures adopted in the first visit to determine the values of VO2max after training. The control group will be performed just one training session total run time conducted in eight sessions by GFP group (approx. 30 min).

ELIGIBILITY:
Inclusion Criteria:

* Strength training practitioner for at least 6 months
* 18 / 45 years
* No injuries

Exclusion Criteria:

* Use of ergogenic resource
* Hypertension and cardiovascular disease
* Drugs

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2016-01; Primary Completion 2016-02 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Oxygen Intake (VO2Max) | Change from Baseline VO2Max after 2 Weeks of Circuit of HIIT

CONTACTS AND LOCATIONS:
Overall Officials: Alberto S. Sá Filho, Dr, Principal Investigator — Iguaçu University